CLINICAL TRIAL: NCT05214053
Title: Cone Beam vs MDCT for Diagnosis and Pre-operative Evaluation of Otosclerosis
Acronym: CONBEAM OTO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: not enough patients
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2021/21
Record Dates: First submitted 2021-12-01; First posted 2022-01-28 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Otosclerosis
Keywords: Otosclerosis; Cone Beam; Conductive hearing loss
MeSH Terms: conditions — Otosclerosis; Hearing Loss, Conductive | interventions — Cone-Beam Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cone Beam CT (Experimental): Each patient will undergo a Cone Beam CT and a MDCT
  Interventions: Device: Cone Beam CT

INTERVENTIONS:
Device: Cone Beam CT — Each patient will undergo a Cone Beam CT and a MDCT

SUMMARY:
This study aims to compare the Cone Beam and the multi-detector computed tomography for diagnosis and pre-operative evaluation of otosclerosis in patients addressed for conductive hearing loss with intact tympanic membrane. The study aims to show that the Cone Beam offers equivalent performances with lower radiation dosage in this indication

DETAILED DESCRIPTION:
Otosclerosis is an inflammatory bone remodeling disorder of the otic capsule, characterized by spongiotic new bone formation, causing stamped ankylosis that can result in conductive hearing loss. Until now, the gold standard imaging technique for diagnosis and pre-operative evaluation of otosclerosis has been multi-detector computed tomography (MDCT). Cone Beam computed tomography is a relatively recent imaging modality. It is associated with a lower radiation dosage compared to MDCT, and a high spatial resolution that allows a more precise analysis of bone structures. During the last 15 years, its use has been increasingly common in odontology and craniofacial surgery. Several studies have already studied the utility of Cone Beam for temporal bone pathologies, including recent retrospective studies that showed satisfying diagnostic performances for otosclerosis. Up to now, very few prospective studies have compared those two imaging modalities for otosclerosis diagnosis and pre-operative evaluation.

Therefore, those two exams will be performed in patients addressed to the hospital for conductive hearing loss with intact tympanic membrane. Thus, the performance of Cone Beam will be compared to MDCT, regarding the positive diagnosis of otosclerosis, the analysis of anatomical structures of the temporal bone for pre-operative evaluation, and also the benefits in terms of irradiation. The MDCTs will include fewer slices than routine MDCTs and will be centered on the area of interest, in order to keep a total radiation dosage smaller or equivalent to routine care

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years and older)
* Requiring radiological assessment for conductive hearing loss with intact tympanic membrane, confirmed by otoscopy and audiogram
* Signed informed consent
* Affiliated or beneficiary of health insurance

Exclusion Criteria:

* Absence of otosclerosis on the MDCT
* History of middle ear surgery
* Pregnancy, breast feeding women and women who are of childbearing age and not practicing adequate birth control
* Patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
False negative rate of Cone Beam for the diagnosis of otosclerosis | 1 day
  False negative rate of Cone Beam for the diagnosis of otosclerosis, compared to MDCT (gold standard).

SECONDARY OUTCOMES:
radiologic grades of otosclerosis | 1 day
  Description of the radiologic grades of otosclerosis, based on Veillon's classification
extension to round window | 1 day
  The parameter that will be assessed is the presence/absence of a bony hypodensity located on the round window bony structure .
  CT will be considered as gold standard. CBCT may be less or equally accurate to detect this small hypodensity area structure
Existence of a bone canal around the labyrinthine portion of the facial nerve | 1 day
  The parameter that will be assessed is the presence /absence of a bony structure covering the VIIth nerve a the level of the oval window.
  CT will be considered as gold standard. CBCT may be less or equally accurate to detect this very thin bony structure , or even better in case of better detection
radiation dosage | 1 day
  Comparison of radiation dosage between Cone Beam and MDCT

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No